CLINICAL TRIAL: NCT01584154
Title: CRYOthermy and Radiofrequency ABLation For AVNRT TrEatment
Brief Title: Comparative Study Between Cryoablation and Radiofrequency Ablation in the Treatment of Supraventricular Tachycardia
Acronym: CRYOABLATE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Ngai Yin Chan, Consultant, Princess Margaret Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1101
Record Dates: First submitted 2012-04-21; First posted 2012-04-24 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Supraventricular Tachycardia; Atrioventricular Nodal Reentrant Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular; Tachycardia, Atrioventricular Nodal Reentry | interventions — Cryosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cryoablation (Experimental)
  Interventions: Procedure: cryoablation
- radiofrequency ablation (Active Comparator): radiofrequency ablation with a 4mm-tip catheter
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: cryoablation — cryoablation with an 8mm-tip catheter
  Arms: cryoablation
Procedure: radiofrequency ablation — radiofrequency ablation with a 4mm-tip catheter
  Arms: radiofrequency ablation

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of cryoablation and radiofrequency ablation in the treatment of the commonest kind of supraventricular tachycardia, namely atrioventricular nodal reentrant tachycardia. The study hypothesis is that cryoablation is non-inferior to radiofrequency.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred for catheter ablation of supraventricular tachycardia and diagnosis of AVNRT is made by cardiac electrophysiology study

Exclusion Criteria:

1. Patients who aged less than 18 or over 80.
2. Patients who are pregnant.
3. Patients who cannot give informed consent.
4. Patients who are judged to have severe mental impairment and cannot report symptoms of palpitation during follow-up.
5. Patients who had previous AVNRT ablation before.
6. Patients who have comorbid congenital heart disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2012-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
treatment success rate, defined as proportion of treated patients with both atrioventricular block-free acute procedural success and mid-term success without recurrence at 6 months | 6 months after treatment

SECONDARY OUTCOMES:
Treatment success rate at 12 months | 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ngai-Yin Chan, MBBS, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Hong Kong, Guangdong, China

REFERENCES:
- [Background] Chan NY, Mok NS, Choy CC, Lau CL, Chu PS, Yuen HC, Lau ST. Treatment of atrioventricular nodal re-entrant tachycardia by cryoablation with an 8-mm-tip catheter versus radiofrequency ablation. J Interv Card Electrophysiol. 2012 Sep;34(3):295-301. doi: 10.1007/s10840-012-9670-9. Epub 2012 Mar 9. PMID 22403042
- [Background] Chan NY, Choy CC, Lau CL, Lo YK, Chu PS, Yuen HC, Choi YC, Lau ST. Cryoablation versus radiofrequency ablation for atrioventricular nodal reentrant tachycardia: patient pain perception and operator stress. Pacing Clin Electrophysiol. 2011 Jan;34(1):2-7. doi: 10.1111/j.1540-8159.2010.02858.x. Epub 2010 Aug 18. PMID 20727096
- [Background] Chan NY, Mok NS, Lau CL, Lo YK, Choy CC, Lau ST, Choi YC. Treatment of atrioventricular nodal re-entrant tachycardia by cryoablation with a 6 mm-tip catheter vs. radiofrequency ablation. Europace. 2009 Aug;11(8):1065-70. doi: 10.1093/europace/eup121. Epub 2009 May 17. PMID 19451097